CLINICAL TRIAL: NCT06351579
Title: A Look at Outcomes After Post Radical Prostatectomy
Brief Title: Data Collection Post Radical Prostatectomy
Acronym: ALTO
Status: Completed | Type: Observational
Sponsor: Levee Medical, Inc. (Industry)
Collaborators: RQM+ (Industry)
Responsible Party: Sponsor
Other Study IDs: 1010159
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence; Radical Prostatectomy; BPH
Keywords: SUI; BPH; Prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Control — This is an observational (registry) study for data collection only. No device or intervention will be used in this study.

SUMMARY:
The study is designed to collect information on patients undergoing radical prostatectomy (RP), with a primary focus on the occurrence, duration, and severity of post-prostatectomy incontinence. Data will be collected at multiple time points, allowing for a dynamic understanding of urinary incontinence patterns at post RP.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is predominantly iatrogenic following radical prostatectomy (RP). Surgical removal of the prostate leads to a shortened urethra, widened bladder neck, and diminished urethral support. This results in increased demand on the urinary sphincter to maintain urinary continence. Most men will experience acute urinary incontinence following RP. Continence progressively improves over time; however, it is estimated that between 5-15% of men will experience chronic urinary incontinence.

Current treatments for post-prostatectomy urinary incontinence include conservative therapies such as pelvic floor muscle training and surgical treatments. The sponsor is conducting a feasibility study (ARID) using a medical device to improve / reduce UI rate at post-RP. This study (ALTO) is designed as a control cohort to collect information on patients undergoing radical prostatectomy (RP) without using the device.

This ALTO study is to systematically collect detailed information on patients undergoing radical prostatectomy, with a primary focus on the occurrence, duration, and severity of post-prostatectomy incontinence. Data will be collected at multiple time points, allowing for a dynamic understanding of urinary incontinence patterns at post RP.

ELIGIBILITY:
Inclusion Criteria:

1. Male 45-70 years of age
2. Diagnosed with prostate cancer and scheduled for radical prostatectomy
3. Gleason Grade Group 3 or lower
4. Prostate size less than 80 grams
5. Able and willing to provide written consent to participate in the study
6. Able and willing to comply with study follow-up visits and procedures

Exclusion Criteria:

1. Malignant tumors outside of the prostate capsule confirmed via baseline assessments (e.g., mpMRI, bone scan)
2. History of urinary incontinence, including stress or urge urinary incontinence
3. On medications to treat overactive bladder (OAB)
4. Presence of urethral stricture or bladder neck contracture
5. Current or chronic urinary tract infection
6. Prior urologic outlet surgical or minimally invasive procedure (e.g., TURP, HoLEP, Rezum, etc.).
7. Prior pelvic radiation or anticipated need for radiation after radical prostatectomy
8. Presence of stones in the bladder
9. History of neurogenic bladder, sphincter abnormalities, or poor detrusor muscle function
10. Body mass index >35
11. History of cancer (excluding prostate cancer meeting the inclusion criteria) which is not considered in complete remission - a potential participant is considered cured if there has been no evidence of cancer within five years of enrollment
12. Diagnosed or suspected primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function, sphincter function or poor detrusor muscle function
13. History of clinically significant congestive heart failure (i.e., New York Heart Association (NYHA) Class III and IV)
14. Insulin-dependent diabetes mellitus
15. Current uncontrolled diabetes (i.e., hemoglobin A1c ≥7.5%)
16. Intravesical prostatic protrusion (IPP) >5mm
17. History of immunosuppressive conditions (e.g., AIDS, post-transplant)
18. Any significant medical history that would pose an unreasonable risk or make the subject unsuitable for the study per investigator discretion
19. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affect the ability to complete the study quality of life questionnaires
20. Subject currently participating in other investigational studies unless approved by the Sponsor in writing

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll male subjects diagnosed with prostate cancer who are scheduled for radical prostatectomy. Subjects must meet all the inclusion criteria and none of the exclusion criteria to participate in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
The change in average 24-hour pad weight over time | Baseline, post-foley, 6 weeks, 3 months, 6 months, and 12 months post-prostatectomy procedure.
  The 24-hour (at-home) pad weight test - The pads are pre-weighed prior to providing them to subjects. The test should be started with an empty bladder. The subject will wear pads and perform their normal daily activities for 24 hours. The subject will be asked to change the pads approximately once every 6 hours during waking hours, or more frequently as needed. The pads will be stored in an air tight bag or container after removal, stored in a refrigerator, and brought to the site at the required follow-up visit for weighing.

SECONDARY OUTCOMES:
Change in pad weight during a 1-hour provocative pad weight test | Baseline, post-foley, 6 weeks, 3 months, 6 months, and 12 months post-prostatectomy procedure.
  The 1-hour pad test involves the following:
  * Subject puts on a pre-weighed pad and is asked to avoid voiding;
  * Subject drinks 500 ml of sodium-free liquid in <15 minutes, then sits or rests;
  * Subjects walks for 30 minutes, including climbing one flight of stairs (up and down)
  * Subject performs the following activities: standing up from sitting (10x), coughing vigorously (10x), running on the spot for 1 minute, bending to pick up an object from the floor (5x), and washing hands in running water for 1 minute;
  * The total amount of urine leaked is determined by weighing the pad. If voiding is urgent and unavoidable, the test is terminated. Collect voiding volume and repeat the test after re-hydration.

OTHER OUTCOMES:
Expanded Prostate Index Composite (EPIC-26) score. | Baseline, post-foley, 6 weeks, 3 months, 6 months, and 12 months post-prostatectomy procedure.
  The Expanded Prostate Cancer Index Composite is a validated, comprehensive questionnaire designed to evaluate patient function and bother after localized prostate cancer treatment. The questionnaire contains 13 items across 5 domains (i.e., urinary incontinence, urinary irritative/obstructive, bowel, sexual and hormonal). Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Choi, Study Chair — Founder and CTO, Levee Medical, Inc
Locations (1):
- LeeveMedical, Inc, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No